CLINICAL TRIAL: NCT00408967
Title: An Open-label Phase II Study of Two Dose Levels of EMD 273066 Administered With Low-dose Cyclophosphamide Following Objective Response to Second-line Chemotherapy in Women With Recurrent Ovarian Carcinoma
Brief Title: Determine if Either of 2 Doses of Study Drug Given With a Low-dose of Cyclophosphamide After a Complete or Partial Response to a Platinum-based Second-line Therapy in Women With Recurrent Ovarian Carcinoma Results in a Longer Time to Progression When Compared to the First Time to Progression.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Th trial got cancelled and no subjects signed informed consent form (ICF); study design not appropriate any longer.
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62206-016
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Ovarian Cancer
Keywords: Ovarian; Cancer; Epithelial; Recurrent; Platinum; Second-line therapy; Maintenance Therapy; Biologic; Targeted Therapy; Antibody
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Recurrence | interventions — tucotuzumab celmoleukin

ARMS (1):
- Tucotuzumab celmoleukin (EMD 273066) (Experimental)
  Interventions: Drug: Tucotuzumab celmoleukin (EMD 273066)

INTERVENTIONS:
Drug: Tucotuzumab celmoleukin (EMD 273066)

SUMMARY:
The purpose of this study is to determine if either of two doses of EMD 273066 when given with a low dose of cyclophosphamide will result in a second time to progression that is as long or longer than the first time to progression

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age 18 years or older
* Have histologically documented ovarian carcinoma (including primary peritoneal carcinoma)
* Have archival tumor tissue available for EpCAM expression determination by immunohistochemistry
* Received first-line platinum-based chemotherapy of up to 8 cycles (approximately 15 to 24 weeks)
* Experienced a complete response to first-line platinum-based chemotherapy
* Experienced a platinum-free interval of at least 6 but not more than 24 months starting at the end of the last cycle of first-line chemotherapy until recurrence

  * Treatment with Avastin (bevacizumab) is permitted during first-line platinum-based chemotherapy through TTP and platinum-based reinduction therapy up to 28 days prior to start of EMD 273066
* Experienced a partial or complete response after up to 8 cycles of second-line platinum-based chemotherapy
* Have a CT/MRI scan within 4 weeks prior to starting treatment
* Be able to start cyclophosphamide and EMD 273066 treatment within 3 to 5 weeks of completion of second-line chemotherapy
* KPS ≥70%
* No clinical history of significantly impaired renal function or chronic kidney disease. Must have an estimated glomerular filtration rate ≥50 mL/min determined by the Cockgroft-Gault-formula
* WBC count ≥2.5x10³/µL (or total granulocytes ≥1x10³/µL)
* Absolute lymphocyte count (ALC) ≥0.5x103/µL
* Platelet count ≥100,000/µL
* Hemoglobin (Hgb) level ≥9 g/dl
* ALT and AST ≤2.5xULN, total bilirubin <1.5xULN
* Serum sodium, potassium and phosphorus within normal limits
* Serum amylase within normal limits
* Serologic testing within 4 weeks prior to starting study treatment with negative results for hepatitis C virus (HCV), human immunodeficiency virus (HIV) and hepatitis B virus (HBV) demonstrated by negative hepatitis B core antibody (HBc Ab) and hepatitis B surface antigen (HbsAg)
* Negative pregnancy test and willingness to use effective contraception for the study duration and 1 month thereafter if of procreative potential

Exclusion Criteria:

* Dyspnea at rest, exercise intolerance
* In any subject with clinically significant non-malignant pulmonary disease: Pulmonary function testing (to include Forced Vital Capacity [FVC] and 1-second Forced Expiratory Volume [FEV-1]) showing <70% of predicted values for FVC or FEV-1 and/or DLCO <50%.
* In any subject with pulmonary or pleural metastatic disease: Arterial oxygen saturation at rest measured transcutaneously on room air < 90% or increased risk for respiratory compromise related to IL2 exposure in the judgment of the investigator.
* ECG with evidence of clinically significant disease within 4 weeks prior to starting study treatment
* Cardiac stress test (e.g., exercise or pharmacological thallium test; exercise or pharmacological echocardiography) with abnormal results within 4 weeks prior to starting treatment in subjects who have a history of coronary heart disease (myocardial infarction, angina pectoris or pathologic coronary angiography)
* Any current evidence of congestive heart failure with NY Heart Association Grade 2 through 4 or echocardiogram with a left ventricular ejection fraction <45% or other signs of clinical significant heart disease
* History of repeated and clinically relevant episodes of syncope or other paroxysmal, ventricular, or other clinically significant arrhythmias
* Evidence of active brain metastases
* Previous malignancy other than ovarian cancer in the last 5 years except basal cell cancer of the skin or pre-invasive cancer of the cervix
* Pregnant or lactating female
* An immediate need for palliative radiotherapy or systemic corticosteroid therapy
* Significant active infection
* Major surgery, chemotherapy, or radiation within 21 days of starting study treatment
* Received another experimental drug within 28 days of starting study treatment
* Uncontrolled hypertension (systolic ≥180 mmHg or diastolic ≥100 mmHg) or hypotension (systolic ≤90 mmHg)
* Presence of medically significant third space fluids such as pleural or pericardial effusions or edema of toxicity grade ≥2 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0 [17].

  * Exception allowed for disease-related peritoneal ascites unless patient requires frequent and repetitive paracentesis management.

Previous diagnosis of an autoimmune disease involving a major organ system

* Transplant recipient on immunosuppressive therapy
* Acute esophageal or gastroduodenal ulcers
* History of prior therapy or a serious uncontrolled medical disorder that in the Investigator's opinion would impair participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12-31 (Actual); Primary Completion 2008-05-31 (Actual); Study Completion 2008-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany